CLINICAL TRIAL: NCT03511287
Title: Effects of Inspiratory Muscle Training in Inspiratory Muscle Function, Functional Capacity, Quality of Life, Lung Function, Breathing Pattern and Thoracoabdominal Motion in Patients With Advanced Lung Disease
Brief Title: Effects of Inspiratory Muscle Training in Patients With Advanced Lung Disease
Acronym: IMTinALD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Veronica Franco Parreira, Full Professor, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNPq 442973/2014-4
Record Dates: First submitted 2018-04-11; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Lung Diseases; Pulmonary Disease
Keywords: inspiratory muscle training; advanced lung disease; maximal inspiratory pressure; inspiratory endurance
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: All patients from the advanced lung disease and pre lung transplantation ambulatory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMT group (Experimental): Group intervention: home-based interval inspiratory muscle training:
  * during 8 weeks (two sessions per day, daily)
  * two times 30 breaths with one-minute rest between them in each session
  * training resistance set to the highest tolerable load according to scores pointed by the patient on the Borg score (between 4 and 6) aiming 50% of actual pimax or higher adjusted in the supervised weekly session
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — Breathing through a device that offers resistance during inspiration. In this study the POWERbreathe device was used (POWERbreathe® K3, HaB International Ltd, UK).

SUMMARY:
The aim of this clinical trial is to evaluate, the effects of inspiratory muscle training program in inspiratory muscle function, functional capacity, quality of life, lung function, breathing pattern and chest wall motion in patients with advanced lung disease. Patients were evaluated before the inspiratory muscle training, after 8 weeks of training and at follow-up which was performed 3 months after the end of the intervention.

DETAILED DESCRIPTION:
Inspiratory Muscle Training (IMT) should be considered an additional intervention in the pulmonary rehabilitation program for patients with advanced lung disease. The aim of this study is to evaluate, the effects of inspiratory muscle training program in inspiratory muscle function, functional capacity, quality of life, lung function, breathing pattern and chest wall motion in patients with advanced lung disease. It is a quasi-experimental study with longitudinal design. Patients with advanced lung disease from the advanced lung disease and pre lung transplantation ambulatory performed home-based high intensity interval IMT for 8 weeks (two sessions per day, daily). In each session patients executed two times 30 breaths with one-minute rest between them. Resistance was set to the highest tolerable according to scores pointed by the patient on the Borg score (between 4 and 6) aiming 50% of actual pimax or higher. An experienced physiotherapist was responsible for weekly adjustments on the resistance of training as well as new assessment of maximal inspiratory pressure. Patients were evaluated before the inspiratory muscle training, after 8 weeks of training and at follow-up which was performed 3 months after the end of the intervention. Patients were evaluated by the same experienced researcher in all three moments of the study. Evaluations were performed in the Laboratory of research and evaluation of cardiorespiratory performance of Federal University of Minas Gerais.

ELIGIBILITY:
Inclusion Criteria:

* presence of inspiratory muscle weakness (Maximal Inspiratory Pressure - MIP ≤ 60 cmH2O or below the reference values proposed for the Brazilian population.
* completion of a 36 sessions of PR or nonattendance in any pulmonary rehabilitation by the time of inclusion and no perspective of initiating it in the next 8 weeks.
* absence of pre-existing neuromuscular, infectious, metabolic, psychiatric diseases or orthopedic problems that prevent from activities of daily living.

Exclusion Criteria:

* presented inspiratory muscle strength higher than 60 cmH2O or predicted value
* unable to follow commands related to the measurements or to the IMT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Inspiratory muscle strength | Before intervention, after 8 weeks intervention and follow-up (3 months after the end of intervention)
  Maximal inspiratory pressure in cmH2O
Change in Inspiratory Muscle Endurance | Before intervention, after 8 weeks intervention and follow-up (3 months after the end of intervention)
  Inspiratory endurance time in seconds

SECONDARY OUTCOMES:
Change in Lung Function | Before intervention, after 8 weeks intervention and follow-up (3 months after the end of intervention)
  Spirometry
Change in Breathing pattern | Before intervention, after 8 weeks intervention and follow-up (3 months after the end of intervention)
  Optoelectronic plethysmography (percentage of contribution of the 3 lung compartments to ventilation)
Change in chest wall motion | Before intervention, after 8 weeks intervention and follow-up (3 months after the end of intervention)
  Optoelectronic plethysmography (lung volumes in liters)
Change in Functional Capacity (direct measure) | Before intervention, after 8 weeks intervention and follow-up (3 months after the end of intervention)
  Six minutes walking distance (meters)
Change in Functional Capacity (inderect measure) | Before intervention, after 8 weeks intervention and follow-up (3 months after the end of intervention)
  London chest activity of daily living scale (total score) - It evaluates the dyspnea in daily activities. Consists in a 15 questions questionnaire with scores from 0-5 in each question. Total score varies from 0 to 75, the higher the score the major the limitation on daily activities due to dyspnea.
Quality of life | Before intervention, after 8 weeks intervention and follow-up (3 months after the end of intervention)
  Saint George Respiratory questionnaire (total score) It is a 50 questions questionnaire. Total score can go from 0 to 100. Higher scores indicate worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Parreira, PhD, Principal Investigator — UFMG
Locations (2):
- Brazil (2):
  - Ambulatório Bias Fortes- Ambulatório de Doença Pulmonar Avançada e Pré Transplante Pulmonar, Belo Horizonte, Minas Gerais
  - Laboratório de Avaliação e Pesquisa em Desempenho Cardiorrespiratório da UFMG, Belo Horizonte, Minas Gerais

IPD SHARING:
Plan to Share IPD: No